CLINICAL TRIAL: NCT07134101
Title: Neoadjuvant Chemoradiotherapy Combined With Serplulimab With or Without Bevacizumab for Locally Advanced Rectal Cancer: A Single-Center, Open-Label, Phase II Randomized Trial
Brief Title: Neoadjuvant Therapy for Locally Advanced Low Rectal Cancer (SMARTi-RC01)
Acronym: SMARTi-RC01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Fu Zan, Director of the Colorectal Cancer Center, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-610
Record Dates: First submitted 2025-08-11; First posted 2025-08-21 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer (Diagnosis)
MeSH Terms: conditions — Colorectal Neoplasms; Disease | interventions — Bevacizumab; Drug Therapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Experimental Arm Induction Phase (2 cycles, every 3 weeks) Chemotherapy: CAPOX (capecitabine + oxaliplatin) or capecitabine monotherapy Capecitabine: 800 mg/m² orally, twice daily (BID), on Days 1-14 of each cycle Oxaliplatin: 130 mg/m² intravenous infusion, on Day 1 of each cycle (if CAPOX) Immunotherapy: Serplulimab 300 mg IV on Day 1 of each cycle Anti-angiogenic therapy: Bevacizumab 5 mg/kg IV on Day 1 of each cycle Radiotherapy: Short-course radiotherapy, 25 Gy in 5 fractions over 1 week Consolidation Phase 2 cycles of CAPOX or capecitabine + serplulimab + bevacizumab Followed by 2 cycles of CAPOX or capecitabine + serplulimab (no bevacizumab) Post-treatment After completion of neoadjuvant treatment, patients will undergo total mesorectal excision (TME) surgery or follow a Watch-and-Wait strategy if a clinical complete response (cCR) is achieved.
  Interventions: Drug: Serplulimab; Drug: Bevacizumab; Radiation: Short-Course Radioterapy; Drug: Chemotherapy (CAPOX or capecitabine)
- Control Arm (Active Comparator): Control Arm Induction Phase (2 cycles, every 3 weeks) Chemotherapy: CAPOX (capecitabine + oxaliplatin) or capecitabine monotherapy Capecitabine: 800 mg/m² orally, twice daily (BID), on Days 1-14 of each cycle Oxaliplatin: 130 mg/m² intravenous infusion, on Day 1 of each cycle (if CAPOX) Immunotherapy: Serplulimab 300 mg IV on Day 1 of each cycle Radiotherapy: Short-course radiotherapy, 25 Gy in 5 fractions over 1 week Consolidation Phase 4 cycles of CAPOX or capecitabine + serplulimab Post-treatment After completion of neoadjuvant treatment, patients will undergo total mesorectal excision (TME) surgery or follow a Watch-and-Wait strategy if a clinical complete response (cCR) is achieved.
  Interventions: Drug: Serplulimab; Radiation: Short-Course Radioterapy; Drug: Chemotherapy (CAPOX or capecitabine)

INTERVENTIONS:
Drug: Serplulimab — Serplulimab 300 mg IV on Day 1
  Other Names: Hanszhuo®
Drug: Bevacizumab — Bevacizumab 5 mg/kg IV on Day 1
  Other Names: Zercepac®
  Arms: Experimental Arm
Radiation: Short-Course Radioterapy — 25 Gy in 5 fractions over 1 week
Drug: Chemotherapy (CAPOX or capecitabine) — Capecitabine: 800 mg/m² orally, twice daily (BID), on Days 1-14 of each cycle Oxaliplatin: 130 mg/m² intravenous infusion, on Day 1 of each cycle

SUMMARY:
The goal of this clinical trial is to learn if combining serplulimab (PD-1 inhibitor) with bevacizumab and short-course total neoadjuvant therapy (TNT) works to treat locally advanced mid-to-low rectal cancer in adults. It will also learn about the safety of this combination.

The main questions it aims to answer are:

Does adding bevacizumab to serplulimab and TNT increase the complete remission rate (cCR + pCR) compared with serplulimab and TNT alone? What medical problems do participants have when receiving these treatments?

Researchers will compare:

Experimental group: serplulimab + bevacizumab + chemotherapy + short-course radiotherapy Control group: serplulimab + chemotherapy + short-course radiotherapy

Participants will:

Receive either the experimental or control regimen for about 4-5 months before surgery or a watch-and-wait approach if complete response is achieved Undergo treatment in cycles that include chemotherapy, immunotherapy (and bevacizumab if in the experimental group), and short-course radiotherapy Visit the clinic regularly for check-ups, blood tests, imaging, endoscopy, and to monitor side effects Be followed for up to 5 years after treatment to assess cancer control, organ preservation, and survival outcomes

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for the study:

1. Age: 18 to 75 years old.
2. Diagnosis: Pathologically confirmed rectal adenocarcinoma with proficient mismatch repair (pMMR) / microsatellite stable (MSS) status, based on biopsy of the primary tumor.
3. Disease Stage: Untreated, preoperative clinical stage cT2-T4 and/or N+, M0 (AJCC 8th edition), unsuitable for initial local excision to achieve radical cure.
4. Tumor Location: Tumor within 8 cm from the anal verge, or assessed by surgeons as not suitable for immediate sphincter-preserving surgery.
5. Organ Preservation Intent: Strong desire for sphincter preservation and willingness to accept close surveillance for at least 2 years after chemoradiotherapy.
6. Surgical Candidacy: Agrees to undergo radical surgery and judged by surgeon to have no contraindication to surgery.
7. Cancer History: No concurrent multiple primary malignancies.
8. Measurable Lesions: At least one measurable or evaluable lesion according to RECIST v1.1 criteria.
9. Life Expectancy: ≥ 3 months.
10. Performance Status: ECOG performance status score of 0-1.
11. Compliance: Good compliance and willingness to sign written informed consent.

Exclusion Criteria:

Participants will be excluded if any of the following conditions apply:

1. Molecular Subtype: Rectal cancer with deficient mismatch repair (dMMR) or microsatellite instability-high (MSI-H) status.
2. Autoimmune Disease: Active, known, or suspected autoimmune disease.
3. Immunodeficiency: Known history of primary immunodeficiency.
4. Transplant History: History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
5. Pregnancy or Lactation: Pregnant or breastfeeding women.
6. Urgent Surgical Indications: Intestinal perforation, gastrointestinal bleeding, or other conditions requiring emergency surgery.
7. Uncontrolled Comorbidities, including but not limited to:

   HIV infection (HIV antibody positive) Active or poorly controlled severe infection Active hepatitis Severe or uncontrolled systemic diseases (e.g., severe psychiatric or neurological disorders, epilepsy, dementia, unstable or decompensated respiratory, cardiovascular, hepatic, or renal disease, uncontrolled hypertension ≥ CTCAE Grade 2 despite medication) Active bleeding or recent thrombotic disease requiring therapeutic anticoagulation, or bleeding tendency, or coagulation abnormalities (INR > 1.5 × ULN, APTT > 1.5 × ULN)
8. Laboratory Abnormalities at Baseline:

   Hemoglobin < 80 g/L Absolute neutrophil count (ANC) < 1.5 × 10⁹/L Platelets < 80 × 10⁹/L ALT or AST > 2.5 × ULN ALP > 2.5 × ULN Total bilirubin ≥ 1.5 × ULN Serum creatinine ≥ 1 × ULN
9. Allergy: Known hypersensitivity to any component of the investigational drugs.
10. Other Clinical Trial Participation: Currently enrolled in another interventional drug clinical trial.
11. Other Conditions: Any other condition judged by the investigator to make the patient unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete Remission (CR) Rate assessed by pathology, MRI, endoscopy, and clinical examination | At the time of surgery for pCR, and at 1 year after achieving cCR for sustained cCR
  Definition: The proportion of participants achieving complete remission, defined as:
  Pathologic complete response (pCR): No residual viable tumor cells detected in the resected specimen after neoadjuvant treatment (ypT0N0) Sustained clinical complete response (cCR): No evidence of residual tumor on digital rectal examination, endoscopy, and MRI, maintained for more than 1 year without surgery Assessment Method: Evaluated by investigators based on imaging, endoscopic findings, pathology (for surgical cases), and clinical examination

SECONDARY OUTCOMES:
Organ Preservation Rate (OPR) assessed by MRI, endoscopy, and clinical examination | From the end of neoadjuvant therapy through 3 years of follow-up.
  Definition: The proportion of participants who achieve organ preservation, defined as avoiding radical rectal resection (TME) without evidence of local tumor recurrence during follow-up.
  Assessment Method: Clinical examination, endoscopy, and MRI.
R0 Resection Rate confirmed by histopathology | At the time of surgery.
  Definition: The proportion of participants who undergo surgical resection with negative microscopic margins (no tumor cells at the resection margin).
  Assessment Method: Pathology review of surgical specimens.
Disease-Free Survival (DFS) measured by imaging and clinical follow-up | Up to 5 years after randomization.
  Definition: Time from randomization to documented disease recurrence (local or distant) or death from any cause, whichever occurs first.
  Assessment Method: Imaging, endoscopic examination, clinical records.
Overall Survival (OS) assessed by survival follow-up | Time Frame: Up to 5 years after randomization.
  Definition: Time from randomization to death from any cause. Assessment Method: Survival status by follow-up visits, phone calls, or registry data.
Objective Response Rate (ORR) assessed by RECIST v1.1 | During neoadjuvant therapy (baseline to pre-surgery evaluation).
  Definition: The proportion of participants achieving a complete response (CR) or partial response (PR) according to RECIST v1.1 during neoadjuvant therapy.
  Assessment Method: MRI, CT scans, and clinical examination.
Disease Control Rate (DCR) assessed by RECIST v1.1 | During neoadjuvant therapy (baseline to pre-surgery evaluation).
  Definition: The proportion of participants achieving CR, PR, or stable disease (SD) as per RECIST v1.1 during neoadjuvant therapy.
  Assessment Method: MRI, CT scans, and clinical examination.
Safety Outcomes assessed by NCI-CTCAE v5.0 | From first dose to 90 days after last dose of study treatment.
  Definition: Incidence, nature, and severity of adverse events (AEs) and serious adverse events (SAEs), graded according to NCI-CTCAE v5.0;

IPD SHARING:
Plan to Share IPD: No